CLINICAL TRIAL: NCT01362023
Title: A Primary-school-based Study to Reduce Prevalence of Childhood Obesity in Terres de l'Ebre (Catalunya (Spain) - EDAL-Educació en Estils Saludables de Vida alimentació-2: Study Protocol for a Randomized Controlled Trial
Brief Title: Efficacy of an Educational School-based Intervention to Reduce Prevalence of Obesity in Childhood-EdAl-2
Acronym: EDAL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: Diputació de Tarragona (Unknown)
Responsible Party: Principal Investigator, Rosa Sola, MD, PhD, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YES
Record Dates: First submitted 2011-05-23; First posted 2011-05-27 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): Control pupils follow their usual activities
- lifestyle counseling (Experimental): In 3 academic years, the intervention program consisted of three components:
  1. Classroom practice by HPA to highlight healthy lifestyle habits
  2. Teaching practice by HPA using books designed to include the nutritional objectives
  3. Parental activities included with their children
  In each of 12 activities (1 h/activity), the classroom practice consisted of three components:
  1. Experimental development of activities regarding each healthy lifestyle habit
  2. Assessment of activity performed in classroom
  3. An activity developed for use at home
  Interventions: Behavioral: lifestyle counseling

INTERVENTIONS:
Behavioral: lifestyle counseling — In 3 academic years, the intervention program consisted of three components:
  1. Classroom practice by HPA to highlight healthy lifestyle habits
  2. Teaching practice by HPA using books designed to include the nutritional objectives
  3. Parental activities included with their children
  In each of 12 activities (1 h/activity), the classroom practice consisted of three components:
  1. Experimental development of activities regarding each healthy lifestyle habit
  2. Assessment of activity performed in classroom
  3. An activity developed for use at home
  Other Names: Childhood obesity
  Arms: lifestyle counseling

SUMMARY:
Our hypothesis is that a regular systematic educational intervention in primary school improves lifestyle choices and reduces obesity. As such, the aim of the study is to evaluate the effects of a 3-year school-based program of lifestyle improvement, including diet and physical activity, implemented by university students acting as "health promoting agents" (HPA) on the prevalence of obesity.

DETAILED DESCRIPTION:
Initial pupil enrollment and continued for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* In the intervention group, all children of the selected classroom are exposed to the intervention.
* The data a will collected on all the children, but only the data from individuals (and their parents) who provided informed consent are included in the final analyses.
* Name, gender, date and place of birth are recorded at the start of the program, while weight, height, body mass index (BMI) and waist circumference variables (identified set of anthropometric measures) are recorded in each of the 3 academic years of the study.

Exclusion Criteria:

* No adequate age
* Lack of inclusion criteria

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Reduction in prevalence of obesity | Changes from baseline in prevalence of obesity at 3 academic years
  Primary outcomes include obesity (BMI ≥95th percentile) and overweight (BMI ≥85th percentile) We will analyzed obesity and overweight and a measure of thinness according to the Cole criteria as well as other measures of adiposity such as BMI z score and waist circumference. The numbers of subjects having a particular dietary habit are expressed as percentages of the total number of individuals being evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Montse Giralt, Md, PhD, Principal Investigator — Universitat Rovira i Virgili, Spain
Locations (1):
- Spain, Amposta, Tarragona, Spain

REFERENCES:
- [Derived] Llaurado E, Tarro L, Morina D, Queral R, Giralt M, Sola R. EdAl-2 (Educacio en Alimentacio) programme: reproducibility of a cluster randomised, interventional, primary-school-based study to induce healthier lifestyle activities in children. BMJ Open. 2014 Nov 20;4(11):e005496. doi: 10.1136/bmjopen-2014-005496. PMID 25412862